CLINICAL TRIAL: NCT03837782
Title: Minimally Invasive Versus Abdominal Radical Resection for Colorectal Cancer
Brief Title: Outcome of Resection for Colorectal Cancer
Acronym: LRLCC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Zhejiang University (Other); Peking University Cancer Hospital & Institute (Other); Zhengzhou University (Other); Peking Union Medical College (Other); Sun Yat-sen University (Other); Fudan University (Other); Shanghai Jiao Tong University School of Medicine (Other); Massachusetts General Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); M.D. Anderson Cancer Center (Other); University of California, Los Angeles (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LRLCC
Record Dates: First submitted 2019-01-31; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Laparoscopy
Keywords: laparoscopy,laparotomy,colorectal cancer
MeSH Terms: interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Intervention Model Description: multicenter, randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients were randomized to be distributed to any group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minimally invasive surgery (Experimental): Patients were randomized to undergo minimally invasive radical resection (endoscopic surgery or robotic assisted surgery). Each participating site required accreditation by the trial management committee to ensure proper surgical technique during minimally invasive surgery.
  Patients were eligible if they had colorectal adenocarcinoma; had a disease stage of I (T1,T2), IIABC (T3-T4ab) or IIIABC (TanyN1-2) according to the staging system of NCCN; and had an Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1 (on a 5-point scale, with higher values indicating greater disability).
  Interventions: Procedure: minimally invasive surgery
- open surgery (No Intervention): Patients were randomized to undergo open radical resection (laparotomy). Each participating site required accreditation by the trial management committee to ensure proper surgical technique during minimally invasive surgery.
  Patients were eligible if they had colorectal adenocarcinoma; had a disease stage of I (T1,T2), IIABC (T3-T4ab) or IIIABC (TanyN1-2) according to the staging system of NCCN; and had an Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1 (on a 5-point scale, with higher values indicating greater disability).
  Exclusion criteria included a history of abdominal or pelvic radiotherapy, or evidence of metastatic disease on positron-emission tomography-computed tomography, magnetic resonance imaging, or computed tomography.

INTERVENTIONS:
Procedure: minimally invasive surgery — Each participating site required accreditation by the trial management committee to ensure proper surgical technique during minimally invasive surgery. No individual surgeons performed only the open approach or only the minimally invasive approach. The committee members reviewed the patients' outcomes and the videos to ensure the adequacy of the surgeon's technique.
  Arms: minimally invasive surgery

SUMMARY:
There are limited data from retrospective studies regarding whether short-term and long-term outcomes after laparoscopic or robot-assisted radical colectomy (minimally invasive surgery) are equivalent to those after open abdominal radical colectomy (open surgery) among patients with early and medium-stage colorectal cancer.

This trial is a multicenter,prospective, randomized trial evaluating short-term and survival outcomes concerning minimally invasive surgery and open surgery for colorectal cancer.

DETAILED DESCRIPTION:
Radical colectomy and proctectomy with regional lymphadenectomy remain the standard recommendation for patients with early and medium-stage colorectal cancer. Current guidelines from the National Comprehensive Cancer Network indicate that either laparotomy (open surgery) or laparoscopy (minimally invasive surgery performed with either conventional or robotic techniques) is an acceptable approach to radical resection in patients with early- and medium stage (I to III) colorectal cancer. These recommendations have led to widespread use of a minimally invasive approach for radical resection, although there is a paucity of adequately powered, prospective, randomized trials evaluating short term and survival outcomes.

Retrospective studies involving patients with early and medium-stage colorectal cancer have shown that laparoscopic resection is associated with less intraoperative blood loss, a shorter length of hospital stay, and a lower risk of postoperative complications than open abdominal radical resection. Similarly, the minimally invasive approach has not been associated with lower 5-year rates of disease-free survival or overall survival than the open approach. In addition, retrospective studies have shown that recurrence rates and survival rates do not differ significantly between the two approaches.

The investigators hypothesized that minimally invasive surgery was not inferior or superior to open radical resection in terms of short-term and long-term outcome. In the present trial, the Laparoscopic Resection and Laparotomy for Colorectal Cancer (LRLCC) Trial, the investigators tested this hypothesis by prospectively assigning patients to minimally invasive (conventional laparoscopic or robotic) or open abdominal radical surgery and comparing the short-term outcome, the rate of recurrence, and the overall survival rate between the two groups.

ELIGIBILITY:
Inclusion Criteria:

(i) tumor without distant metastasis; (ii) classified as stage I, II or III by TNM staging system; (iii) Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1; (iv) a minimum of 12 lymph nodes resected to accurately identify stage; (v) solitary malignant lesion after thorough colonoscopy; (vi) complete resection (R0) with no positive nodes left behind; (vii) histological diagnosis of adenocarcinoma.

Exclusion Criteria:

(i) <18 years or >90 years; (ii) serious concurrent illness; (iii) clinically suspicious distant metastasis detected by positron emission tomography-computed tomography (PET-CT); (iv) familial adenomatous polyposis syndrome (FAP), hereditary non-polyposis colorectal cancer (HNPCC) and other hereditary CRC; (v) postoperative pathological close, indeterminate, or positive margins; (vi) circumferential resection margin < 1mm in rectal cancer; (vii) short anticipated life expectancy due to postoperative comorbidities on account of cardiopulmonary insufficiency.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
complications | through hospital stay, an average of two weeks
  complications includes intraoperative and postoperative complications, such as huge blood loss, anastomotic fistula, abdominal infection and septic shock.
disease free survival | From date of randomization until the date of first documented progression, assessed up to 70 months
  Disease-free survival (DFS) was defined as the interval between the date of surgical resection and diagnosis of recurrence or the most recent follow-up date.
overall survival | From date of randomization until the date of death from any cause, assessed up to 70 months.
  Overall survival (OS) was measured from the date of hepatectomy to death with or without HCC recurrence or the end of this study period.

CONTACTS AND LOCATIONS:
Overall Officials: Dalu M Kong, M.D., Study Director — Tianjin Medical University
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China